CLINICAL TRIAL: NCT03098069
Title: Kangaroo Mother Care Implementation Research for Accelerating Scale-up
Brief Title: Implementation Research on Scaling up Kangaroo Mother Care (KMC)
Acronym: KMC-Scaleup
Status: Completed | Type: Observational
Sponsor: Society for Applied Studies (Other)
Collaborators: Government of Haryana (Unknown); All India Institute of Medical Sciences (Other); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: ERC.0002716
Record Dates: First submitted 2017-03-16; First posted 2017-03-31 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2018-04

CONDITIONS: Low Birth Weight Babies; Kangaroo Mother Care Scale up
Keywords: Kangaroo Mother Care; Low Birth Weight; Implementation research

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KMC Scale up in a district: This is an implementation research project on scaling up KMC in selected government and private health facilities in an entire district, aiming to cover newborns weighing less than 2000gms at birth.

SUMMARY:
This implementation research aims to accelerate effective and high coverage of Kangaroo Mother Care in district Sonipat in the state of Haryana, India. The project is being led by government of Haryana. KMC units will be set up in selected government and private delivery facilities. KMC will be initiated for all babies with birth weight less than 2000 gm in the facilities (either in born or referred from elsewhere) and continued at home post discharge. These babies may be either born in the facility or referred to the facility. A linkage with community health workers will be established to support mothers to continue KMC at home.

DETAILED DESCRIPTION:
Babies born with low birth weight are at increased risk of mortality. The global burden of low birth weight babies is high with 15 million neonates being born preterm each year. Complications from preterm births result in over one million deaths, comprising 35% of all newborn mortality.

The way forward is to achieve an effective and equitable implementation of all those interventions for which evidence of efficacy is well established. One of the efficacious interventions is Kangaroo Mother Care (KMC). KMC has been demonstrated to promote physiologic stability, facilitate early breastfeeding, provide a thermally supportive environment, reduce the risk of serious infections, and reduce the mortality of hospitalized, stable preterm and low birth weight infants. This practice also promotes bonding between infants and their mothers during the first hours and days of life. The "Every Newborn Action Plan" endorsed and launched by the World Health Assembly in May 2014 includes the goal of scaling up KMC to 50% of babies weighing under 2000 grams by 2020, and to 75% of these babies by 2025.

This implementation research aims to promote KMC scale up in a district of Haryana. The steps include formative research to identify barriers and facilitators; designing of scalable models to deliver KMC across the facility-community continuum; implementation and evaluation of these models aiming towards wider national or state-level scale-up. Learning at each stage of this process will be applied to refining and improving the KMC delivery model. This proposal aims to develop, implement and evaluate a delivery model for KMC. The study will be implemented in two phases: i) development of a delivery model and ii) implementation and evaluation of the model.

The performance of the model will be assessed against a pre-defined success criterion of 80% or higher coverage of effective KMC at the population level.

KMC will be implemented at three levels, pre-facility, facility and post-facility.

ELIGIBILITY:
Inclusion Criteria:

* Babies with birth weight less than 2000g born in the study area.

Exclusion Criteria:

* Newborns who are severely sick will have the initiation of KMC delayed until stabilization.

Ages: 1 Minute to 28 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study participants will include babies of birth weight less than 2000g born in the study area. Newborns who are severely sick according to pre-defined criteria will have the initiation of KMC delayed until they have stabilized.
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Effective coverage of KMC at discharge from hospital | At the time of discharge from hospital, will vary with each baby
  Proportion of babies who weighed less than 2000g at birth and got KMC for atleast 8 hours and were exclusively breastfed in the last 24 hours, assessed at discharge.
Effective coverage of KMC at home, 7 days after hospital discharge | 7 days after discharge from hospital
  Proportion of babies who weighed less than 2000g at birth and got KMC for atleast 8 hours and were exclusively breastfed in the last 24 hours, assessed at 7 days after hospital discharge.

SECONDARY OUTCOMES:
Population-level duration of KMC | First 28 days of life
  Number of days KMC was received by infants in the population with birth weight less than 2000gm during the neonatal period.
Any KMC received | First 28 days of life
  Percent of infants with birth weight less than 2000gm receiving any KMC i.e. any duration in last 24 hours, at 28 days of life
Infants exclusively breastfed | First 28 days of life
  Percent of infants with birth weight less than 2000gm exclusively breastfed in the last 24 hours, ascertained at discharge, 7 days post discharge and 28 days of life
Neonatal mortality | 1 year
  Number of deaths in infants between birth to 28 days of life expressed per 1000 live births.
Cost of KMC scale up | 1 year
  Cost estimation of establishing KMC units in selected delivery facilities, recurring cost of implementing KMC in these units and cost of implementing KMC at home post discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Sarmila Mazumder, MBBS, PhD, Principal Investigator — CHRD, Society for Applied Studies
Locations (1):
- CHRD, Society for Applied Studies, Sonīpat, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mony PK, Tadele H, Gobezayehu AG, Chan GJ, Kumar A, Mazumder S, Beyene SA, Jayanna K, Kassa DH, Mohammed HA, Estifanos AS, Kumar P, Jadaun AS, Hailu Abay T, Washington M, W/Gebriel F, Alamineh L, Fikre A, Kumar A, Trikha S, Ashebir Gebregizabher F, Kar A, Bilal SM, Belew ML, Debere MK, Krishna R, Dalpath SK, Amare SY, Mohan HL, Brune T, Sibley LM, Tariku A, Sahu A, Kumar T, Hadush MY, Gowda PD, Aziz K, Duguma D, Singh PK, Darmstadt GL, Agarwal R, Gebremariam DS, Martines J, Portela A, Jaiswal HV, Bahl R, Rao Pn S, Tadesse BT, Cranmer JN, Hailemariam D, Kumar V, Bhandari N, Medhanyie AA; KMC Scale-Up Study Group. Scaling up Kangaroo Mother Care in Ethiopia and India: a multi-site implementation research study. BMJ Glob Health. 2021 Sep;6(9):e005905. doi: 10.1136/bmjgh-2021-005905. PMID 34518203
- [Derived] Medhanyie AA, Alemu H, Asefa A, Beyene SA, Gebregizabher FA, Aziz K, Bhandari N, Beyene H, Brune T, Chan G, Cranmer JN, Darmstadt G, Duguma D, Fikre A, Andualem BG, Gobezayehu AG, Mariam DH, Abay TH, Mohan HL, Jadaun A, Jayanna K, Kajal FNU, Kar A, Krishna R, Kumar A, Kumar V, Madhur TK, Belew ML, M R, Martines J, Mazumder S, Amin H, Mony PK, Muleta M, Pileggi-Castro C, Pn Rao S, Estifanos AS, Sibley LM, Singhal N, Tadele H, Tariku A, Lemango ET, Tadesse BT, Upadhyay R, Worku B, Hadush MY, Bahl R; KMC Scale-Up Study Group. Kangaroo Mother Care implementation research to develop models for accelerating scale-up in India and Ethiopia: study protocol for an adequacy evaluation. BMJ Open. 2019 Nov 21;9(11):e025879. doi: 10.1136/bmjopen-2018-025879. PMID 31753865